CLINICAL TRIAL: NCT03551652
Title: Evaluation of Duration of Curarisation (Surgical Efficacy) and Pharmacokinetics of Neuromuscular Block After a Single Dose of Rocuronium in Geriatric Patients (Age ≥ 80 Years ) Compared to a Younger Population (Age < 50 Years).
Brief Title: Comparison of Duration of Neuromuscular Block in Geriatric Patients Compared to Young Patients.
Acronym: NMB-old-age
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: NMB-old-age
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2020-11

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Young patients: Patients aged 18 - 50 years
  Interventions: Drug: Pharmacokinetics of rocuronium induced neuromuscular block
- Geriatric patients: Patients aged ≥ 80 years
  Interventions: Drug: Pharmacokinetics of rocuronium induced neuromuscular block

INTERVENTIONS:
Drug: Pharmacokinetics of rocuronium induced neuromuscular block — Measurement of rocuronium induced neuromuscular block comparing patients aged > 80 years with patients aged 18 to 50 years

SUMMARY:
Elderly people, especially geriatric patients, account for a growing share of patients receiving anesthesia.

In patients over 75 years of age the annual rate of anesthesia represents 16.8 / 100 inhabitants for women and 19.6 / 100 for men. It is a growing population, but also the most fragile population with a mortality amounting to 44.4 / 10000 anesthesia. After 85 years, one out of every two patients is ASA 3 or older.

The first cause of death related to anesthesia today remains respiratory complications, particularly infectious.

This is a major public health issue right now. The studies on the use of curare and particularly rocuronium are old and did not study a population of elderly people (with an average age of 70 years). Several studies show an increase in the duration of neuromuscular blockade in patients older than 70 years irrespective of any renal failure, with sometimes persistent curarizations more than 2h after a single dose. But no study to date has studied the duration of deep-intensity neuromuscular block (TOF).

DETAILED DESCRIPTION:
Scientific justification Elderly patients, especially geriatric patients, represent an increasing percentage of patients receiving anesthesia. Thus, among the population over 75 years old, the annual rate of anesthesia represents 16.8 / 100 inhabitants. women and 19.6 / 100 in men. This is a growing population, but also the most fragile population with a mortality amounting to 44.4 / 10000 anesthesia. After 85 years, one out of every two anesthetized patients is ASA 3 or higher. The first cause of mortality linked to anesthesia today remains respiratory complications, particularly those of infectious origin. The care of this population presents a major public health challenge. Studies on the use of curare and especially rocuronium are relatively old and did not study a geriatric population, so in the group aged the average age was 70 years.

Several studies show an increase in the duration of neuromuscular blockade in patients over the age of 70, regardless of any renal failure, with extremes of persistent curarization more than 2 h after a single dose. However, no study to date has investigated the duration of deep-tissue neuromuscular blocking (train of four (TOF) <1) required for performing certain surgical procedures, including laparoscopic surgery.

Several studies show that elderly patients have increased sensitivity to residual curarization.

In this context, a study on the kinetics of the curare and in particular rocuronium is necessary in order to evaluate if the "standard" induction dose of 0.6 mg / kg is adapted to this population or if this dose requires an adjustment to reduce the respiratory risks associated with residual curarization.

General description of the research Objectives To compare the duration of curarization induced by rocuronium (0.6 mg / kg of real weight) between young patients (18-50 years old) and old men (> 80 years old).

Evaluation criteria

Primary judgment criterion:

Total curarization time (DCT, defined as the sum of the installation time + deep curarization time + recovery time The installation time (Dinstall) is defined as the time between the injection of rocuronium and the disappearance of the responses to the train of four (TOF = 0).

The deep block duration (Dprof) is defined as the time between the disappearance of the responses to the train of four (TOF = 0) and the reappearance of the first response to a train of four (TOF = 1).

The recovery time (Drécup) will be evaluated for both a T4 / T1 recovery ≥ 0.9 (Drécup0.9) and a T4 / T1 ratio ≥ 1.0 (Drécup1.0). recovery will also be assessed by the ratio of T4/Tref, i.e. the ratio of the 4th response to a TOF stimulation and the mean of the 4 responses to a TOF stimulation before administration of a neuromuscular blocking agent. This ratio is measured by the TofScan (IdMed, Marseille, France).

Research Methodology Patients will be anesthetized, as in clinical routine, with propofol in target controlled infusion anesthesia (TCI) according to the Schnider model at the effect site. Analgesia will be provided either by remifentanil or sufentanil.

Neuromuscular block will be monitored using TofScan (IdMed, Marseille, France), with accelerometry measurement at the adductor pollicis. The TOF-WatchSX will be calibrated in cal 2 mode, as defined by the manufacturer. (12) Neuromuscular blockade will be induced by a single dose of rocuronium 0.6 mg / kg of actual weight. The intensity of the neuromuscular block will be measured by a train of four every 15 s from the curare injection to TOF = 0 (Dinstall): then every minute until TOF = 1 (Dprof); then every minute until T4/T1 ≥ 0.9 (Drécup0.9) and T4/T1 ≥ 1.0 (Drécup1.0). Dinstall, Dprof, Drécup0.9 and Drécup1.0 will be recorded, as well as time to recovery of T4/Tref of 0.9 and 1.0.

Patient selection: inclusion and non-inclusion criteria, recruitment modality

Criteria for inclusion:

* Patient aged 18 to 50 or ≥ 80 years
* Body mass index (BMI) between 18.5 and 35
* Intervention requiring general anesthesia with intubation

Criteria of non-inclusion:

* Rocuronium allergy
* Need for rapid sequence induction
* Clinically apparent hepatocellular insufficiency
* Renal insufficiency requiring dialysis
* ASA> 2 in the group of 18 to 50 years

Materials and techniques used Monitoring of the TofScan (IdMed, Marseille, France) monitor at the level of the adductor pollicis. The electrodes are placed at the ulnar edge of the arm 2 cm apart.12 Registration of the Tref value before administration of rocuronium. Measurement of the neuromuscular block intensity every 15s from the neuromuscular blocking facility to TOF = 0, then measured every minute of the neuromuscular block up to TOF = 1(Dprof) and finally measured every minute until decurarisation spontaneous T4 / T1 ≥ 0.9 (Drécup0.9) and T4 / T1 ≥ 1.0 (Trécup1.0). The time to recovery of T4/Tref to 0.9 and 1.0 ill also be recorded.

Normothermia is maintained (temperature> 36 ° C) by the use of a forced air system (Bair Hugger) with temperature monitoring by oesophageal probe.

Statistics

Number of patients:

To estimate the number of patients to be included in each group, we postulate that the DCT of patients 80 and over is, on average, at least 30% greater than the CSD of patients under 50 years of age.

The mean DCT of the under-50 group is around 60 minutes and a standard deviation of 11 minutes. By setting the alpha risk at 5% and the expected power 80%, it will be necessary to include 14 patients per group, or 28 in total.

Statistical analysis :

Descriptive analysis: calculation of%, means, standard deviations, quartiles and extreme values Principal analysis: the mean DCT will be compared by a matched series average comparison test, then by a linear regression model with adjustment for potential confounders, excluding matching factors.

Secondary analyzes: The secondary endpoints will be compared by a MacNémar test and a Student's t-test on matched series and possibly by conditional logistic and linear regression models to allow an adjustment for potential confounding factors.

Threshold of significance: 5% Software: SAS v9.4

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery with neuromuscular blockade by rocuronium
* Body mass index between 18.5 and 35
* Age 18 - 50 years or age > 80 years

Exclusion Criteria:

* Known allergy to rocuronium
* rapid sequence induction
* clinical hepatocellular insufficiency
* renal insufficiency requiring dialysis
* ASA class > 2 in the group 18-50 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged between 18-50 years or > 80 years, undergoing surgery with neuromuscular block induced by rocuronium
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Total time of neuromuscular block | 4 hours, during surgery
  Time from rocuronium injection to total recovery of neuromuscular block

SECONDARY OUTCOMES:
Deep neuromuscular block | 4 hours, during surgery
  Time between TOF=0 and TOF=1
Recovery time 0.9 | 4 hours, during surgery
  Time between TOF=0 and T4/T1≥0.9
Recovery time 1.0 | 4 hours, during surgery
  Time between TOF=0 and T4/T1≥1.0
Recovery time 0.9 Tref | 4 hours, during surgery
  Time between TOF=0 and T4/Tref≥0.9
Recovery time 1.0 Tref | 4 hours, during surgery
  Time between TOF=0 and T4/Tref≥1.0

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fuchs-Buder, MD, PhD, Principal Investigator — CHRU de Nancy
Locations (1):
- CHRU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klopfenstein CE, Herrmann FR, Michel JP, Clergue F, Forster A. The influence of an aging surgical population on the anesthesia workload: a ten-year survey. Anesth Analg. 1998 Jun;86(6):1165-70. doi: 10.1097/00000539-199806000-00005. PMID 9620497
- [Background] Auroy Y, Laxenaire MC, Clergue F, Pequignot F, Jougla E, Lienhart A. [Anesthetics according to characteristics of patients, establishments and indications]. Ann Fr Anesth Reanim. 1998;17(11):1311-6. doi: 10.1016/s0750-7658(99)80043-4. No abstract available. French. PMID 9972358
- [Background] Forrest JB, Rehder K, Cahalan MK, Goldsmith CH. Multicenter study of general anesthesia. III. Predictors of severe perioperative adverse outcomes. Anesthesiology. 1992 Jan;76(1):3-15. doi: 10.1097/00000542-199201000-00002. PMID 1729933
- [Background] Pignaton W, Braz JRC, Kusano PS, Modolo MP, de Carvalho LR, Braz MG, Braz LG. Perioperative and Anesthesia-Related Mortality: An 8-Year Observational Survey From a Tertiary Teaching Hospital. Medicine (Baltimore). 2016 Jan;95(2):e2208. doi: 10.1097/MD.0000000000002208. PMID 26765400
- [Background] Tiret L, Desmonts JM, Hatton F, Vourc'h G. Complications associated with anaesthesia--a prospective survey in France. Can Anaesth Soc J. 1986 May;33(3 Pt 1):336-44. doi: 10.1007/BF03010747. PMID 3719435
- [Background] Yamamoto H, Uchida T, Yamamoto Y, Ito Y, Makita K. Retrospective analysis of spontaneous recovery from neuromuscular blockade produced by empirical use of rocuronium. J Anesth. 2011 Dec;25(6):845-9. doi: 10.1007/s00540-011-1229-x. Epub 2011 Sep 21. PMID 21935686
- [Background] Comparison of Neuromuscular Blockade with Rocuronium in Young and Elderly Patients with or without Renal Failure. 1SK Gvalani, 2L Pradeep Research & Innovation in Anesthesia, July-December 2016;1(2):45-51
- [Background] Bevan DR, Fiset P, Balendran P, Law-Min JC, Ratcliffe A, Donati F. Pharmacodynamic behaviour of rocuronium in the elderly. Can J Anaesth. 1993 Feb;40(2):127-32. doi: 10.1007/BF03011309. PMID 8443851
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear TD, Vender JS, Parikh KN, Patel SS, Patel A. Residual Neuromuscular Block in the Elderly: Incidence and Clinical Implications. Anesthesiology. 2015 Dec;123(6):1322-36. doi: 10.1097/ALN.0000000000000865. PMID 26448469
- [Background] Arain SR, Kern S, Ficke DJ, Ebert TJ. Variability of duration of action of neuromuscular-blocking drugs in elderly patients. Acta Anaesthesiol Scand. 2005 Mar;49(3):312-5. doi: 10.1111/j.1399-6576.2005.00634.x. PMID 15752394
- [Background] Kocabas S, Yedicocuklu D, Askar FZ. The neuromuscular effects of 0.6 mg kg(-1) rocuronium in elderly and young adults with or without renal failure. Eur J Anaesthesiol. 2008 Nov;25(11):940-6. doi: 10.1017/S0265021508004717. Epub 2008 Jun 9. PMID 18538050
- [Background] Neuromuskuläres Monitoring in Klinik und Forschung. T. Fuchs-Buder, Springer Medezin Verlag, 2008, ISBN 978-3-540-78569-9
- [Derived] Schmartz D, Sghaier R, Bernard P, Fils JF, Fuchs-Buder T. Neuromuscular block in patients 80 years and older: a prospective, controlled study. BMC Anesthesiol. 2021 Sep 13;21(1):225. doi: 10.1186/s12871-021-01443-1. PMID 34517841